CLINICAL TRIAL: NCT04981470
Title: A First in Human Study of Feasibility of Baroloop: The Baroloop Study
Brief Title: The Baroloop Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Device modifications needed
Sponsor: neuroloop GmbH (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL_CIP-FIH
Record Dates: First submitted 2021-07-20; First posted 2021-07-29 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Investigational Device (Experimental): Subjects implanted with the baroloop device
  Interventions: Device: baroloop System

INTERVENTIONS:
Device: baroloop System — vagal nerve stimulation

SUMMARY:
The baroloop Study is a non-randomized, prospective, single-arm, multi center First in Human (FIH) study with the primary objective being the assessment of the safety and feasibility of using the baroloop System in subjects with uncontrollable hypertension. The secondary objective is to document the effect of the baroloop device on the blood pressure and quality of life in subjects with hypertension. Up to 10 subjects will be enrolled in up to 3 sites in Europe.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older and less than 80 years of age.
2. Persistent office systolic blood pressure (SBP) ≥ 140 mm Hg and diastolic blood pressure (DBP) > 90 mm Hg on antihypertensive medicines on two visits separated by a minimum of four weeks.
3. Mean 24-hour systolic ABPM ≥ 130 mm Hg and mean 24 hour diastolic ABPM ≥ 80 mm Hg conducted after direct observed therapy to confirm that antihypertensive medicines were taken as prescribed during the ABPM measurement.
4. Stable drug regimen of 4 antihypertensive medicines consisting of a renin-angiotensin blocker(ACE) or Angiotensin II Receptor Blocker (ARBs), a calcium channel blocker (CCB), a diuretic and spironolactone for 4 weeks at treatment. If spironolactone is not tolerated, the regimen must include instead the addition of further diuretic therapy with either eplerenone, amiloride, higher-dose thiazide/thiazide-like diuretic or a loop diuretic, or the addition of bisoprolol or doxazosin. If none of these medicines are tolerated, then patients on a 3-drug regimen may be included.
5. The Investigator has confirmed that the patient has already tried and/or is not suitable for treatment with currently CE-marked device-based therapies for resistant hypertension as an alternative to baroloop therapy.
6. Willingness and ability to comply with follow-up requirements.
7. Signed informed consent.

Exclusion Criteria:

1. Any patient in whom access to the vagal nerve is limited by the size of the vagus (a size not compatible with the baroloop cuff).
2. Any patient with a history of injury to the vagus nerve or its branches (e.g., the recurrent laryngeal nerve).
3. Secondary causes of hypertension.
4. Calculated eGFR < 30 mL/min/1.73m2.
5. Type 1 diabetes mellitus or poorly controlled type 2 diabetes mellitus (HbA1c > 10%).
6. One or more episodes of orthostatic hypotension in the past year
7. Requirement for chronic oxygen therapy or mechanical ventilation.
8. Untreated (no CPAP therapy) sleep apnea (AHI > 15)
9. Morbid obesity, defined as Body Mass Index >40 kg/m2 or arm circumference 46 cm.
10. Pacemaker and/or implantable defibrillators.
11. History of transient ischemic accident or cerebrovascular accident during six (6) months prior to screening.
12. Symptomatic carotid artery disease or > 70% occlusion of either carotid artery; any carotid malformation or lesion, a carotid bruit or other abnormal carotid sound.
13. Prior surgery, radiation therapy or scarring in the neck in the region of the carotid artery (e.g., patients with a tracheostomy, extensive thymectomy or thyroid surgery).
14. Limited mobility of the neck secondary to vertebral disease or prior vertebral surgery, including patients who wear a cervical support.
15. History of heart failure (NYHA class III-IV or ejection fraction < 30%), myocardial infarction, unstable angina, coronary bypass or coronary angioplasty during six (6) months prior to screening.
16. Cardiac arrythmias (atrial fibrillation, atrial flutter, etc.) that require anticoagulation or interfere with a consistent measurement of blood pressure.
17. Syncope in the last 6 months.
18. History of bleeding disorders, thrombocytopenia, hemophilia or significant anemia (hemoglobin (Hgb) < 10 gm/dl).
19. Current anticoagulation therapy (excluding antiplatelet therapy with aspirin as a sole therapy).
20. Works night shifts.
21. History of unresolved drug or alcohol use.
22. Active treatment of a psychiatric ailment.
23. Life expectancy of less than 12 months due to other disease.
24. Subject has a condition that, in the opinion of the investigator, precludes participation, including willingness to comply, with all follow-up procedures.
25. Participation in another clinical study for which follow-up is currently on-going.
26. Women who are of child-bearing age or who have the potential to become pregnant
27. Resting heart rate of <40 beats/min for patients on beta blockers or <60 beats/min for all other patients, confirmed at both baseline visits.
28. Baroreflex failure or autonomic neuropathy
29. Symptomatic, uncontrolled bradyarrhythmias
30. Atrioventricular block of any grade
31. Patients who are treated with Pacemaker and/or implantable defibrillators
32. Presence of a vagus stimulator
33. Patients who expect to require magnetic resonance imaging (MRI) of the cervical area
34. Occupational exposure to high levels of non-ionizing radiation that may interfere with therapy
35. Patients with a limited ability to read, understand and execute adjustment procedures (for example, persons suffering from dementia).
36. Likely exposure to diathermy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wilko Spiering, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Investigational Device
Started | 4
Completed | 0
Not Completed | 4
Not completed — Device failure in all 4 patients | 4

BASELINE CHARACTERISTICS:
Arm/Group | Investigational Device
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Netherlands | 4

OUTCOME MEASURES:

1. Primary Outcome: Composite Major Adverse Event (MAE) Rate
Description: The MAE rate is calculated based on the number of participants that either died, were hospitalized for hypertensive crisis after the first titration visit, or experienced any device or procedure-related serious adverse events.
Time Frame: at 6 months post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device
Number analyzed (Participants) | 4
Participants | 4

2. Primary Outcome: Feasibility - Device Placement and Vagal Nerve Stimulation
Description: Feasibility was calculated based on the number of participants in whom the baroloop system was successfully placed around a vagal nerve and stimulation of the nerve was possible. Stimulation of the vagus nerve was attempted for the first time after either 14 or 21 days; depending on the healing progress of the participant after the surgery. Therefore, feasibility (ability to place the device and ability to stimulate the nerve after the surgery) was either confirmed after 14 days or 21 days, depending on the healing progress of the participant after the surgery.
Time Frame: Day 14 or Day 21 post-implantation
Measure: Count of Participants; unit: Participants
Arm/Group | Investigational Device
Number analyzed (Participants) | 4
Participants | 4

3. Secondary Outcome: Change in Blood Pressure
Description: Change in blood pressure recorded during intraoperative stimulation
Time Frame: at the time of implantation
Reporting Status: Not Posted

4. Secondary Outcome: Change in 24-hour ABPM
Description: Mean change of 24-hour ambulatory systolic and diastolic blood pressure post-treatment versus baseline
Time Frame: 1, 3, 6, 12, 18 and 24 months
Reporting Status: Not Posted

5. Secondary Outcome: Composite MAE Rate
Description: he MAE consists of all causes of death, hospitalization for hypertensive crisis post-titration, and any device or procedure-related serious adverse events
Time Frame: 1, 3, 12, 18 and 24 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in Office Blood Pressure
Description: Mean change in office systolic and diastolic blood pressure
Time Frame: 1, 3, 6, 12, 18 and 24 months
Reporting Status: Not Posted

7. Secondary Outcome: Change in Antihypertensive Drugs/Dosages
Description: Changes in antihypertensive drugs/dosages post-implantation as analyzed by Daily Defined Dosages (WHO Definition) and total medications
Time Frame: 1, 3, 6, 12, 18 and 24 months
Reporting Status: Not Posted

8. Secondary Outcome: Quality of Life Evaluation - Short Form (36) Health Survey
Description: Quality of Life as measured by the Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36). The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Time Frame: Baseline, 1, 3, 6, 12, 18 and 24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for each patient until he or she left the study. As all patients exited the study due to device failure, the period of time AEs were collected varies from 95 to up to 598 days.
Arm/Group | Investigational Device
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 4/4
Other Adverse Events (participants affected / at risk) | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=4)
explantation surgery due to device failure (Surgical and medical procedures) | 4 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigational Device (N=4)
Dizziness after charging the device (General disorders) | 1 (1)
Pressure on larynx (General disorders) | 1 (1)
Reddening around chest wound after implant procedure (Surgical and medical procedures) | 1 (1)
Abscess left groin (Infections and infestations) | 1 (1)
Heart palpitations after medication increase (Cardiac disorders) | 2 (2)
Dizziness (General disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Dyspnea occurred after discontinuation of furosemide
Covid 19 infection (Infections and infestations) | 1 (1)
Bursitis in left shoulder (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest pain, sensation of sickness, dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/70/NCT04981470/Prot_SAP_000.pdf